CLINICAL TRIAL: NCT06402149
Title: Comparison of 2 Different Methods in Infraclavicular Block
Status: Enrolling by invitation | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E1-23-3323
Record Dates: First submitted 2023-04-13; First posted 2024-05-07 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Pain; Nerve Block; Analgesics
Keywords: infraclavicular block; VAS (Visual Analogue Scale) score; dexamethasone
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grup I: Patients who underwent infraclavicular block by lateral sagittal method under USG guidance by adding 2ml dexamethasone (8mg) 3cc 0.9% NaCl to local anesthetic containing 10 ml of bupivacaine (0.5%) and 5cc of prilocaine (2%) will be included in Group I.
  Interventions: Other: dexamethasone
- Grup II: Patients who underwent infraclavicular block by lateral sagittal method under USG guidance by adding 10 ml of bupivacaine (0.5%) and 5ml of prilocaine (2%) and 5 cc of 0.9% NaCl will be included in Group II.

INTERVENTIONS:
Other: dexamethasone — Use of dexamethasone in infraclavicular block
  Other Names: infraclavicular block
  Groups: Grup I

SUMMARY:
Background :The investigators wanted to see if dexamethasone, which is routinely used as an adjuvant tool by different anesthesiologists in the orthopedics operating room, can really start the effect of other local anesthetics early and prolong the duration of action during infraclavicular block, and giving less additional analgesics after surgery.

Aims:The investigators plan to determine whether this outcome of , dexamethasone which is routinely used as an adjuvant tool to prolong postoperative analgesia.

Methods :60 participants will be included in the study. It includes participants the age of 18, who do not have lung disease such as COPD (Chronic Obstructive Pulmonary Disease), who will undergo infraclavicular block, and who are mentally healthy with ASA I-III.After obtaining written consent from the premedication unit from the participants who were preoperatively evaluated, a vascular access will be opened in the non-operated arm and 0.09% NaCl will be started and 0.05 mg/kg midazolam will be given. All patients will be monitored. With nasal cannula, 3lt/min O2 will be started. 3lt/min O2 will be started with nasal cannula. Patients who underwent infraclavicular block by lateral sagittal method under USG(ultrasound) guidance by adding 2ml dexamethasone (8mg) 3cc 0.9% NaCl to local anesthetic containing 10 ml of bupivacaine (0.5%) and 5cc of prilocaine (2%) will be included in Group I. Patients who underwent infraclavicular block by lateral sagittal method by adding 10 ml of Bupivacaine (0.5%) and 5ml of prilocaine (2%) and 5 cc of 0.9% NaCl will be included in Group II.

ASA score of the patients, drugs used in surgery, name of surgery, age, weight, height, block time, surgery start and end time, pre-block vitals, post-block vitals, adverse effects, sensory and motor block scale, with 10-minute intervals after the block, after the operation. grades immediately after, 12 hours and 24 hours, VAS scoring at 12 and 24 hours after surgery, surgeon satisfaction will be recorded. In addition, morphine and other analgesic consumption will be checked in all patients in the first 24 hours after surgery.

DETAILED DESCRIPTION:
Background : The investigators to see if dexamethasone, which is routinely used as an adjuvant tool by different anesthesiologists in the orthopedics operating room, can really start the effect of other local anesthetics early and prolong the duration of action during infraclavicular block, thus enabling the surgery to start early and giving less additional analgesics after surgery.

Aims:The investigators plan to determine whether this outcome of dexamethasone , which is routinely used as an adjuvant tool to prolong postoperative analgesia.

Methods :60 participants will be included in the study. It includes participants over the age of 18, who do not have lung disease such as COPD (Chronic Obstructive Pulmonary Disease), who will undergo infraclavicular block, and who are mentally healthy with ASA I-III.After obtaining written consent from the premedication unit from the participants were preoperatively evaluated, a vascular access will be opened in the non-operated arm and 0.09% NaCl will be started and 0.05 mg/kg midazolam will be given. All participants will be monitored. With nasal cannula, 3lt/min O2 will be started. 3lt/min O2 will be started with nasal cannula. Participants who underwent infraclavicular block lateral sagittal method under USG guidance by adding 2ml dexamethasone (8mg) 3cc 0.9% NaCl to local anesthetic containing 10 ml of bupivacaine (0.5%) and 5cc of prilocaine (2%) will be included in Group I. Participants underwent infraclavicular block by lateral sagittal method by adding 10 ml of Bupivacaine (0.5%) and 5ml of prilocaine (2%) and 5 cc of 0.9% NaCl will be included in Group II.

ASA score of the participants, drugs used in surgery, name of surgery, age, weight, height, block time, surgery start and end time, pre-block vitals, post-block vitals, adverse effects, sensory and motor block scale, with 10-minute intervals after the block, after the operation. grades immediately after, 12 hours and 24 hours, VAS (Visual Analogue Scale) scoring at 12 and 24 hours after surgery, surgeon satisfaction will be recorded.In addition, morphine and other analgesic consumption will be checked in all patients in the first 24 hours after surgery.

At the end of the study, statistical analysis will be made parametrically and non-parametrically through the SPSS 2021 program. Statistics consultancy will be taken when necessary.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patient group who will undergo upper extremity surgery will be included in the study.

Exclusion Criteria:

* Patients under the age of 18 who have lung diseases that will prevent blocking and who are not mentally healthy will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients will be included in the study. It includes patients over the age of 18, who do not have lung disease such as COPD, who will undergo infraclavicular block, and who are mentally healthy with ASA I-III.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-08-10 (Estimated); Study Completion 2024-08-16 (Estimated)

PRIMARY OUTCOMES:
Analgesia duration | 24 hours
  A comparison will be made in both groups by looking at the sensory block onset time and the time between the patient's first analgesia request.

SECONDARY OUTCOMES:
Morphine other analgesics consumption | 24 hours
  The morphine and other analgesics consumption will be measured in all patients in the first 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Esma M Simsek, M.D., Principal Investigator — Ankara City Hospital Bilkent; Hülya Kaşıkara, M.D., Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gouda N, Zangrilli J, Voskerijian A, Wang ML, Beredjiklian PK, Rivlin M. Safety and Duration of Low-Dose Adjuvant Dexamethasone in Regional Anesthesia for Upper Extremity Surgery: A Prospective, Randomized, Controlled Blinded Study. Hand (N Y). 2022 Nov;17(6):1236-1241. doi: 10.1177/15589447211008558. Epub 2021 Apr 21. PMID 33880959
- [Background] Pehora C, Pearson AM, Kaushal A, Crawford MW, Johnston B. Dexamethasone as an adjuvant to peripheral nerve block. Cochrane Database Syst Rev. 2017 Nov 9;11(11):CD011770. doi: 10.1002/14651858.CD011770.pub2. PMID 29121400
- [Derived] Simsek EM, Kasikara H. Dexamethasone Added to Mixed Local Anesthetics in Infraclavicular Block: The Dexamethasone Paradox in Chronic Pain. Niger J Clin Pract. 2025 Aug 1;28(8):955-961. doi: 10.4103/njcp.njcp_36_25. Epub 2025 Aug 30. PMID 40884325
- See also: pubmed — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9608287/
- See also: pubmed — https://pubmed.ncbi.nlm.nih.gov/29121400/